CLINICAL TRIAL: NCT02020213
Title: Effectiveness of Posaconazole as Salvage Treatment After 2 Weeks of Preemptive Antifungal Treatment
Brief Title: Posaconazole as Salvage Therapy for Aspergillus Pulmonary Infection.
Acronym: Posaconazole
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF13263
Record Dates: First submitted 2013-12-05; First posted 2013-12-24 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Clinical Infection
Keywords: successful percentage
MeSH Terms: conditions — Communicable Diseases | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posaconazole, salvage (Other): Posaconazole, per oral , 400 mg, bid , 8 weeks.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — 400 mg po bid for 8 weeks
  Other Names: posanol

SUMMARY:
Invasive Aspergillus infection (IAI) occasionally occurs in immunocompromised people. Except administrating empirical anti-fungal agent, using objective parameters to support the tentative diagnosis of an IAI in order to make the anti-fungal treatment more specifically is also important. At present, serum galactomannan (GM) test is the less-invasive, non-cultural, and time-saving examination for augmenting a diagnosis of Aspergillosis. It was suggested by Infectious Disease Society of America (IDSA) 2008 as a screening and monitoring tool for Aspergillosis , and the cut-off value was adjusted to 0.5 by USA FDA . However, in clinical practice, GM seems not to have good predicted value even the sensitivity and specificity are declaimed more than 80% . Other controversial issues include the reproducibility of GM5 and the effect of piperacillin-tazobactam or other antibiotics on the accuracy of GM baseline In this study, serum GMs are examined in two conditions, one is collected for establishing a baseline and the other is collected after piperacillin-tazobactam administration. We hope to confirm the validity of GM baseline and the effect of piperacillin-tazobactam on GM value in Taiwan.

DETAILED DESCRIPTION:
We try to enroll patient who are followed in hematology department in TCVGH and are diagnosed as probable pulmonary Aspergillus infection or proven pulmonary Aspergillus infection. If they have poor response to current thought effective agent for pulmonary Aspergillus (eg, amphotericin B, Voriconazole, itraconazole) 2 weeks, then they can choose to receive Posaconazole as salvage therapy in our study. However, our study wants to quantification of therapeutic response, so the enrolled patient should be agree to let us check serum galactomannan level at beginning and per 2 weeks. They also should be receive chest CT in the beginning and in the end of posaconazole treatment. The rule out timing is evaluated by clinical doctors (hematology department) per 2 weeks, if posaconazole has poor effect to their disease, the clinical doctors can decided to terminate posaconazole administration. Another effective agent will be given when posaconazole fails.

ELIGIBILITY:
Inclusion Criteria:

* Taichung Veterans General Hospital Hematology and Oncology patients with pulmonary aspergillosis, the preliminary use of effective anti-Aspergillus drugs (including amphotericin B, itraconazole, or voriconazole) 14 days later, the symptoms worsen or improve, or can not tolerate the side effects.
* The default number of subjects 12.

Exclusion Criteria:

* Children, minors, pregnant women, newborns, prisoners, mental illness, loss of adult decision-making capacity due to illness, the Aboriginal ... and other vulnerable groups, and critically ill patients

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
clinical response | per 2 weeks
  fever subsides (< 38 C) dyspnea improves ( evaluate by clinical doctors) CXR improves

SECONDARY OUTCOMES:
serum galactomannan level | per 2 weeks
  follow the galactomannan level and check if it corresponds to clinical response or not.

CONTACTS AND LOCATIONS:
Overall Officials: Sz-Rung Huang, Bachelar, Study Director — Chief of Infection department,TCVGH Pu-Li branch